CLINICAL TRIAL: NCT03851042
Title: Use of Virtual Reality for Postoperative Pain After Laparoscopic Hysterectomy
Brief Title: Virtual Reality for Postoperative Pain After Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Nichole Mahnert, Nichole Mahnert, MD, Associate Professor Dept of Obstetrics and Gynecology, MIS Fellowship Co-Director, Endometriosis and Chronic Pelvic Pain Clinic, UofA, BUMCP, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1806640289
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: patients will be randomized to either receive virtual reality headsets in the post anesthesia recovery unit (PACU) as an adjunct therapy or undergo routine postoperative management.
Who Masked: Participant
Masking Description: Upon enrollment, the patient will be randomized using the REDcap randomization tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Virtual Reality Head set in PACU (Experimental): Use of VR Headset in PACU post hysterectomy for up to 4 hours.
  Interventions: Device: Virtual Reality Head set in PACU
- No intervention (Active Comparator): Routine PACU care post hysterectomy for up to 4 hours
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Virtual Reality Head set in PACU — Use of VR headset to determine post op satisfaction in PACU, decreased pain reduction and opioid consumption
  Arms: Virtual Reality Head set in PACU
Other: No intervention — Routine post laparoscopic hysterectomy management (no VR headset)
  Arms: No intervention

SUMMARY:
Patients will be randomized to either receive virtual reality headsets in the post anesthesia recovery unit (PACU) as an adjunct therapy or undergo routine postoperative management. Pain scores will be recorded at standardized intervals in the PACU. The patient will be asked to complete a survey at their two week post op visit assessing their satisfaction with their post op recovery.

The purpose of this study is to determine whether a virtual reality relaxation program used in the immediate postoperative period after laparoscopic hysterectomy will decrease pain scores and reduce both oral and intravenous opioid consumption.

DETAILED DESCRIPTION:
According to the CDC, 115 Americans die every day due to opioid overdose. Prescription opioid related overdose deaths accounted for 40% of all opioid deaths in the US in 2016. In surgery, opioids are an effective tool in reducing pain in the postoperative state. However, this may lead to dependence if pain control is poorly managed. A study examining analgesic use after low risk surgery found that patients requiring a second prescription for opioids within 7 days of their surgery were 44% more likely to become long-term opioid users one year after their surgery.

n order to combat this issue, the concept of multi-modal analgesia has been promoted to reduce the use of opioids for postoperative pain. This modality includes medications (e.g. NSAIDS), regional anesthesia, and adjunct therapies such as meditation and acupuncture.

Virtual reality (VR) is an emerging technology in which a person is immersed in an environment through visual and audio cues that effect the senses. These effects can lead to all types of reactions based on the content and as such, virtual reality is used as a platform for, amongst other things, entertainment, education and patient care.

In health care, virtual reality has been used to desensitize patients with various phobias, provide surgical training and as an effective tool for pain control. At this time, there are no studies demonstrating the use of virtual reality for pain control after gynecologic surgery.

This is a feasibility study to asses if VR can be used for postoperative pain control and whether a VR relaxation program used in the immediate post operative period after laparoscopic hysterectomy will decrease pain scores and reduce both oral and intravenous opioid consumption. If this study is feasible the investigators would then be able to perform a larger study, which could show if VR does or does not reduce postoperative pain. Possible benefits from this study include improved pain control requiring less narcotic medications during the time spent in the PACU after laparoscopic hysterectomy for benign indication. It could also provide improvement of anxiety associated with the postoperative period. This intervention could be a benefit for all women who desire to use non-pharmacologic measures for pain control during the immediate postoperative period. Alternatively, the patient can proceed without the intervention if desired. There are many other pain control methods that the patient can still use during the study. Nothing will be withheld from the patient due to the study.

Recruitment will take place in the outpatient clinic and the preoperative area of the Main Operating Room or Same Day Surgery Once a potential study patient has been identified, a written informed consent form will be provided by a member of the research team to the patient. The member of the team will review the consent form with the patient and she will have the opportunity then to chose to voluntarily participate or decline with the understanding, should she decline, this will in no way affect her care. After all her questions have been answered and she elects to participate in the study, she will sign the consent and a signed copy of the consent will be provided to her for her records. This will be at not cost to the subjects.

Risks include exacerbation of claustrophobia, anxiety, nausea, vomiting due to how the VR works. There are very few risks associated with the intervention. There is a 0.025% risk of seizures, particularly in patients with a known seizure disorder. Theoretically patients with claustrophobia could have exacerbated symptoms, however, these symptoms have not been seen and recorded. Patients with these risk factors will be excluded from the study. There is another theoretical risk of increased nausea, although this has not been shown to occur in previous studies site them.

Our exclusion criteria helps to reduce the possibility of adverse effects from experiencing VR. Once consent forms are signed, they will be kept in a locked drawer of the fellow involved. All data will be collected via RED cap, which is a secure website. When the patient is randomized, they will be given a subject number. This will be used to de-identify the patient.

Adverse events/reactions will be reported to the UA IRB. In the case of injury or illness resulting from this study, emergency medical treatment is available from Banner University Medical Center Phoenix but will be provided at the usual charge. No funds have been set aside to compensate the participant in the event of injury. Their insurance company will be charged for continuing medical care and/or hospitalization.

To assure their study-related costs are paid for, all study-related procedures/tests must be conducted at a Banner Health facility.

he data collection sheets will be stored in the fellows office (Room 3113, 1441 N 12th St. Phoenix, AZ 85006). Information from these forms, and demographic data collected from the patient's chart will be stored in REDcap and only be accessible by members of the study.

Subjects can decide to be removed from the study at any time from when they first consent to the study to when they fill out the survey at the two week postoperative visit. Their withdrawal will be noted in RED cap. The paper forms used to collect data will be destroyed and their virtual data collection sheets will be deleted from REDCap.

All consents will be done in either private exam rooms within the Women's Institute clinic in the 1441 Building of Banner University Medical Center or the private preoperative bay on the day of surgery. Only those involved in consenting and data collection will be allowed to access the consent forms and place data in REDCap.

The patient would be committed to the study during the postoperative recovery period in the PACU, which is approximately 4 hours. They will also be asked to complete a brief survey at the time of their 2 week postoperative visit. If not, they will be mailed the survey to complete and return.

The control group will have no changes to routine PACU protocol. They will be asked to rate their pain at defined intervals that can later be compared to the pain scores of the intervention group. Morphine equivalents during PACU stay will be calculated for the control group. The intervention group will also be offered the routine PACU protocol. The only change being the addition of offering the VR intervention which includes the Samsung VR Innovator edition goggle set, fitted with Samsung Galaxy Note 4 mobile phone. The module options are provided from Applied VR and include Guided relaxation (30 minutes), a tour of Iceland (3 minutes), Dream Beach (30 minutes), Dolphin Swim (15 minutes), Farm Sanctuary (5 minutes), Seal Hospital (10 minutes), and Wild West (5 minutes).

Prior to each new subject use, fabric surfaces of the Samsung Gear set will be cleaned with VIrex, Sani-Wipes will be used to clean the plastic housing, and the glass lenses will be cleaned with an alcohol-based lens cleaner. Each headset will be fitted with a sanitary disposable fabric cover on the VR goggles for new users. Each subject will also wear fitted head caps that minimize direct contact with the devices. At time of recruitment, patients will be given the opportunity to try on the VR goggles and watch the four chosen VR modules that will be offered during their PACU recovery period. At that time, subjects will be instructed on how to apply the head gear. Subjects will apply and remove the headgear themselves, while their trained PACU nurses will be able to assist them in adjusting head straps once the VR goggles have been placed. Subjects will be able to discontinue use of the VR goggles at any time they wish, including before the conclusion of their chosen VR module. There is no minimum or maximum amount of time patients will be allotted to participate in VR modules during their PACU stay. The total amount of time using the VR system and number of separate uses will be recorded. After each patient completes the study, the disposable head cap, fabric covers and foam backing from the devices will be discarded.

It is routine for patients to follow up two weeks after their surgery for a postoperative visit. At that time, they will be asked to complete a survey addressing their satisfaction with the postoperative recovery process in the PACU. If they are not seen in 2 weeks, the survey will be mailed, or the subjects will be contacted via phone to complete the survey.

Up to 30 patients will be recruited for this pilot study. A Master Log will be created that includes patient ID number, patient name, MRN, and date of surgery. The data collection form will be created that includes patient ID number, age, height, weight, BMI, VR Y/N, preoperative diagnosis, past medical history, ASA classification, initial pain score, final pain score, total morphine equivalents used during post-anesthesia recovery unit (PACU) stay, length of time from admission to discharge from PACU, number of uses of VR, total VR use time, and other medications given also include if/when local analgesic was used, what type and where. RedCap is an online data tool that will be used as to collect and store data. At the end of the study, the Master Log, which will be the only document containing patient identifiers will be destroyed.

A review of the study will be performed half way through the process (when 15 subjects have participated) to assess the safety of the study. The investigators will assess how many, if any, of the participants in the study had adverse effects to the protocol.

It is estimated that this study will take 6 months to complete, and therefore around the 3 month mark or at 15 subjects (whichever comes first) will be the point at which a preliminary safety study will be done by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing laparoscopic hysterectomy
* Benign indications
* Dr. Jamal Mourad or Dr. Nichole Mahnert will be performing hysterectomy

Exclusion Criteria:

* Non-English speakers
* History of chronic opioid use
* History of epilepsy
* History of claustrophobia
* Have received a prescription or taken opioids within 2 weeks for their scheduled surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
PACU satisfaction survey | 2 weeks post operative visit
  Survey asking questions regarding their satisfaction with use of VR. A 7-point Likert scale will be used to assess satisfaction with VR modality. 1- very dissatisfied, 2-disatisfied, 3-neutral, 4-satisfied, 5-very satisfied
Meds used at home post op for pain control | 2 week postoperative op visit
  Patients will be asked about specific medications used at home for post op pain control. We will specifically determine the morphine equivalents used for opioids.
Visual Analogue scale for pain | Immediately following surgery
  This is a 1-10 scale that will be asked to patients to assess pain level while in the postoperative care unit, 0=no pain on a graduated scale to 10=worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Foley, MD, Study Director — Director Department of Obstetrics and Gynecology BUMCP
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDC Opioid Overdose. (August 30, 2017). Retrieved from https://www.cdc.gov/drugoverdose/epidemic/index.html
- [Background] Alam A, Gomes T, Zheng H, Mamdani MM, Juurlink DN, Bell CM. Long-term analgesic use after low-risk surgery: a retrospective cohort study. Arch Intern Med. 2012 Mar 12;172(5):425-30. doi: 10.1001/archinternmed.2011.1827. PMID 22412106
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Aman MM, Jason Yong R, Kaye AD, Urman RD. Evidence-Based Non-Pharmacological Therapies for Fibromyalgia. Curr Pain Headache Rep. 2018 Apr 4;22(5):33. doi: 10.1007/s11916-018-0688-2. PMID 29619620
- [Background] Triscari MT, Faraci P, Catalisano D, D'Angelo V, Urso V. Effectiveness of cognitive behavioral therapy integrated with systematic desensitization, cognitive behavioral therapy combined with eye movement desensitization and reprocessing therapy, and cognitive behavioral therapy combined with virtual reality exposure therapy methods in the treatment of flight anxiety: a randomized trial. Neuropsychiatr Dis Treat. 2015 Oct 7;11:2591-8. doi: 10.2147/NDT.S93401. eCollection 2015. PMID 26504391
- [Background] Yiannakopoulou E, Nikiteas N, Perrea D, Tsigris C. Virtual reality simulators and training in laparoscopic surgery. Int J Surg. 2015 Jan;13:60-64. doi: 10.1016/j.ijsu.2014.11.014. Epub 2014 Nov 18. PMID 25463761
- [Background] Schmitt YS, Hoffman HG, Blough DK, Patterson DR, Jensen MP, Soltani M, Carrougher GJ, Nakamura D, Sharar SR. A randomized, controlled trial of immersive virtual reality analgesia, during physical therapy for pediatric burns. Burns. 2011 Feb;37(1):61-8. doi: 10.1016/j.burns.2010.07.007. Epub 2010 Aug 7. PMID 20692769